CLINICAL TRIAL: NCT00875758
Title: Phase II Study of Late- Versus Early Treatment of Post-hemorrhagic Ventricular Dilation in Preterm Infants.
Brief Title: Optimizing Treatment of Post-hemorrhagic Ventricular Dilation in Preterm Infants
Acronym: LETAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LETAP-09-0380
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Intraventricular Hemorrhage; Hydrocephalus
Keywords: preterm infants; IVH; germinal matrix; intraventricular hemorrhage; hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard threshold (Active Comparator)
  Interventions: Procedure: Removal of CSF through ventricular access device
- Low-threshold (Experimental)
  Interventions: Procedure: Removal of CSF through a ventricular access device

INTERVENTIONS:
Procedure: Removal of CSF through ventricular access device — Ventricular access devices (VADs) are surgically implanted when cranial ultrasound measures reach treatment group-specific criteria. For the standard-threshold arm, VADs will be implanted when the age-adjusted ventricular index shows the ventricles to be at the 97th percentile + 2 standard deviations. Cerebrospinal fluid is then removed from the VADs 1-3 times daily as required to maintain ventricles within these parameters.
  Arms: Standard threshold
Procedure: Removal of CSF through a ventricular access device — Ventricular access devices (VADs) are surgically implanted when cranial ultrasound measures reach treatment group-specific criteria. For the standard-threshold arm, VADs will be implanted when the age-adjusted ventricular index shows the ventricles to be at the 97th percentile. Cerebrospinal fluid is then removed from the VADs 1-3 times daily as required to maintain ventricles within these parameters.
  Arms: Low-threshold

SUMMARY:
Intraventricular hemorrhage remains the most frequent, severe neurological complication of prematurity, occurring in 25-30% of preterm infants. Post-hemorrhagic ventricular dilation (PHVD) occurs in 25-50% of those infants, with over half requiring ventriculoperitoneal shunts. When suboptimally untreated, PVHD results in a 3-4 fold increase in neurodevelopmental delay. Despite the lifelong impact of PHVD on quality of life, little research has been done over the past 20 years to improve patient outcomes.

The CENTRAL HYPOTHESIS of this project is that early treatment of PHVD will reduce shunt-dependence and improve neurodevelopmental outcome in preterm infants.

DETAILED DESCRIPTION:
Cranial ultrasound (CUS) is routinely performed on preterm infants ≤ 34 weeks estimated gestational age (EGA) on day-of-life (DOL) #3 and again on DOL #7-10. Patients with Papile Grade II-IV intraventricular hemorrhage (IVH) will undergo serial CUS 1-3 times weekly for 21 days following IVH to monitor for post-hemorrhagic ventricular dilation (PHVD). Using standardized CUS parameters (Levene's ventricular index, Davies's diagonal anterior horn width and thalamo-occipital diameter), infants will be offered enrollment in the trial when their ventricular measures exceed the 97th percentile. Randomization to either low- or standard-threshold PHVD treatment will be performed by opening sequentially numbered, sealed envelopes. Envelopes will be prepared using a randomization schedule where allocations are assigned in a 1:1 ratio in blocks of 4 so that the desired 1:1 ratio will be maintained at periodic intervals in the study.

Neurosurgical treatment of progressive PHVD involves surgical placement of a ventricular access device (VAD) for the removal of cerebrospinal fluid (CSF). Though at present clear criteria do not exist for CSF removal, an estimation of usual neurosurgical practice and that used in previous trials (standard-threshold) is intervention at Levene's EGA-adjusted 97th percentile for ventricular enlargement + 4 mm or greater (> 2 standard deviations > 97th percentile) or a diagonal width enlargement of the frontal horn > 10 mm. For the purpose of this study, low-threshold intervention will be defined as ventricular enlargement > 97th percentile with either a frontal diagonal width 7-10 mm or a thalamo-occipital diameter >24 mm.

CUS will be performed 2-3 times weekly in both the low- and standard-threshold groups. CSF will be removed under sterile conditions via VAD taps (10 ml/kg over 20 minutes, 0-4 times daily) as needed to maintain the CUS ventricular dimensions defined above for each treatment group. Treatment group-specific ventricular size must be achieved within 48-72 hours of VAD placement, and ventricles must be maintained within this range throughout the duration of treatment.

If CSF removal is still required at 44 weeks EGA and there is consensus among the treating neonatologist and neurosurgeon, permanent VP shunts will be surgically implanted. The rate of VP shunts required by 44 weeks EGA and by 12 months corrected age will be monitored. Formal neurodevelopmental evaluations will be performed by a blinded developmental psychologist at 18-24 months corrected age to assess neurocognitive and psychomotor function in low- versus standard-threshold groups. Each infant will be scored using the Bayley Scales of Infant Development.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at ≤ 34 weeks estimated gestational age with ultrasound-confirmed IVH will be followed for eligibility.
* All infants with any grade IVH will be carefully followed with serial ultrasounds 1-3 times weekly to monitor ventricular measures.
* All infants with any grade IVH will be carefully followed for their ventricular measures. If ventricular measures are crossing percentile lines toward the 90th then the infant will be considered for recruitment as soon as the measures cross 97th.

Exclusion Criteria:

* Infants with congenital cerebral malformations
* Cystic periventricular leukomalacia
* CNS infection, metabolic disease
* PHVD present at birth will be excluded from the study.

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2009-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Ventriculoperitoneal shunt-dependence | One year

SECONDARY OUTCOMES:
Shunt malfunction | 4 years
Unnecessary device implantation | One year
Shunt infection | One year
Neurodevelopmental Outcome | 18-24 months of age

CONTACTS AND LOCATIONS:
Overall Officials: David D Limbrick, MD, PhD, Principal Investigator — Washington University School of Medicine; Amit Mathur, MD, Principal Investigator — Washington University School of Medicine; Terrie Inder, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] de Vries LS, Liem KD, van Dijk K, Smit BJ, Sie L, Rademaker KJ, Gavilanes AW; Dutch Working Group of Neonatal Neurology. Early versus late treatment of posthaemorrhagic ventricular dilatation: results of a retrospective study from five neonatal intensive care units in The Netherlands. Acta Paediatr. 2002;91(2):212-7. doi: 10.1080/080352502317285234. PMID 11952011
- [Background] Brouwer A, Groenendaal F, van Haastert IL, Rademaker K, Hanlo P, de Vries L. Neurodevelopmental outcome of preterm infants with severe intraventricular hemorrhage and therapy for post-hemorrhagic ventricular dilatation. J Pediatr. 2008 May;152(5):648-54. doi: 10.1016/j.jpeds.2007.10.005. Epub 2007 Dec 26. PMID 18410767